CLINICAL TRIAL: NCT03415438
Title: Assessment of Thoracolumbar Fascia Length in Patients With Subacromial Impingement Syndrome
Brief Title: Assessment of Thoracolumbar Fascia Length
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Professor, Baskent University
Other Study IDs: KA17/273
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Fascia
Keywords: thoracolumbar fascia; subacromial impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Assessments will be done for 30 patients diagnosed as subacromial impingement syndrome in physical medicine and rehabilitation department of Baskent University.
  Interventions: Diagnostic Test: Visual Analogue Scale; Diagnostic Test: posterior capsule tightness; Diagnostic Test: shortness tests for lumbar movements; Diagnostic Test: range of motion tests for lumbar movements; Diagnostic Test: The thoracolumbar fascia length test; Diagnostic Test: Modify Schober test
- Group 2: Assessments will be done for 30 healthy volunteers
  Interventions: Diagnostic Test: Visual Analogue Scale; Diagnostic Test: posterior capsule tightness; Diagnostic Test: shortness tests for lumbar movements; Diagnostic Test: range of motion tests for lumbar movements; Diagnostic Test: The thoracolumbar fascia length test; Diagnostic Test: Modify Schober test

INTERVENTIONS:
Diagnostic Test: Visual Analogue Scale — intensity of pain perception patients feel
Diagnostic Test: posterior capsule tightness — tape measurement for posterior capsule tightness with patients lying at side and horizontally adducting their shoulder.
Diagnostic Test: shortness tests for lumbar movements — tape measurement for lumbar movements
Diagnostic Test: range of motion tests for lumbar movements — range of motion measurements for lumbar flexion, extension and lateral flexion with goniometer.
Diagnostic Test: The thoracolumbar fascia length test — patient sitting straight with shoulders at horizontal plane, both the arms are asked to rotated with primarily spinal rotation. the degree of rotation gives idea about the thoracolumbar fascia length
Diagnostic Test: Modify Schober test — tape measurement of spinal flexion between designated regions

SUMMARY:
The purpose of the study is to compare the elasticity of thoracolumbar fascia in patients with and without subacromial impingement syndrome.

30 patients diagnosed as subacromial impingement syndrome in physical medicine and rehabilitation department of Baskent University will be recruited as group 1. 30 healthy volunteers will be recruited as group 2. Visual Analogue Scale (VAS) with the aim of assessing pain severity, tape measurement for posterior capsule shortness; body lateral flexion, rotation and extensor movements and lumbar extensor shortness will be observed for correlation with thoracalumbal fascia flexibility. Lateral flexion, flexion, and extension movements will be measured using goniometry for trunk normal joint movements. The thoracolumbar fascia length test and Modify Schober test will be used for thoracolumbar fascia length.

ELIGIBILITY:
Inclusion Criteria:

* 30 patients with Subacromial Impingement Syndrome and 30 volunteers
* between ages of 20-40 years
* both sexes

Exclusion Criteria:

* having lumbar surgery
* having problem with lumbar region in last 6 months
* having scoliosis
* radiologically diagnosed kiphosis
* MR diagnosed lumbar and thoracic herniation
* positive sacroiliac tests
* restricted pelvic motion
* having scapular dyskinesia

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 patients with Subacromial Impingement Syndrome and 30 volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
thoracolumbar fascia length test | 1 week
  thoracolumbar fascia length

SECONDARY OUTCOMES:
Visual Analogue Scale measurement in cm with 0 pointing no pain and 10 pointing worst pain. patient marks the intensity of his/her pain in a 10 cm line and researcher measures the intensity of the pain with a tape. | 1 week
  pain intensity
Goniometric measurement | 1 week
  lumbar movements
Shortness measurement with tape measurement in cm. patient stretches the posterior capsule and the beginning and the end positions are measured with tape. | 1 week
  posterior capsule shortness
lumbar extensor shortness test measurement in cm | 1 week
  lumbar extensor shortness

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided